CLINICAL TRIAL: NCT00992771
Title: A Pilot, Randomized, Double-blind, Placebo-controlled Phase I Study to Determine the Safety and Tolerability of Varenicline (Chantix®) in Treating Spinocerebellar Ataxia Type 3
Brief Title: Study to Determine the Safety and Tolerability of Varenicline (Chantix®) in Treating Spinocerebellar Ataxia Type 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Ataxia Foundation (Other); Bob Allison Ataxia Research Center (BAARC) (Unknown); Pfizer (Industry)
Responsible Party: Principal Investigator, Theresa Zesiewicz, Professor of Neurology, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Spinocerebellar Ataxia Type 3
MeSH Terms: conditions — Machado-Joseph Disease | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Varneicline (Experimental)
  Interventions: Drug: varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — up to 1mg BID for 8 weeks
  Arms: Varneicline
Drug: placebo — placebo matching varenicline, up to 1mg BID for 8 weeks
  Arms: Placebo

SUMMARY:
Spinocerebellar ataxia (SCA) is a group of inherited disorders characterized by cerebellar degeneration leading to imbalance, incoordination, speech difficulties and problems with walking. Recently, individual case reports have suggested that varenicline, a drug used in smoking cessation, produces substantial improvement in patients with several inherited ataxias. A modest response was noted in 5 patients with SCA, suggesting that it is potentially efficacious in this disorder as well. Although this agent is available for off-label use, the severe side effects noted with its use and the lack of long-term toxicity data demand that it be systematically assessed. The present study will test whether varenicline is safe and potentially efficacious in a heterogeneous cohort of adults with SCA.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with spinocerebellar ataxia type 3 diagnosed by a movement disorder specialist and confirmed by genetic testing (of the patient or in a first degree relative of the patient).
2. Age 18 years to 80 years.
3. Women of child-bearing potential must use a reliable method of contraception and must provide a negative pregnancy test at entry into the study.
4. Serum creatine kinase, complete metabolic panel, complete blood count, liver function tests, renal function tests, platelets and EKG are within normal limits (results obtained from primary care physician and dated within the past 6 months or obtained at screening visit).
5. Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
6. Ability to ambulate with or without assistance.
7. Score of 10 or higher (worse) on the SARA total score.
8. Score of 3 or higher (worse) on the 'gait' subsection of the SARA rating scale.

Exclusion Criteria:

1. Any unstable illness or concomitant medical condition that, in the investigator's opinion, precludes participation in this study. This includes other disorders that may affect gait or balance (stroke, arthritis, etc).
2. Pregnancy or lactation.
3. Concurrent participation in another clinical study.
4. Patients with a history of substance abuse.
5. Patients who currently smoke or have smoked within the past 12 months.
6. Presence of psychosis, bipolar disorder, untreated depression (BDI greater than or equal to 21), or history of suicide attempt.
7. Concurrent treatment with any MAOIs, Wellbutrin, or nicotine patches.
8. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini Mental Status Exam score less than 24).
9. Legal incapacity or limited legal capacity.
10. Presence of severe renal disease (BUN 50% greater than normal or creatinine clearance <60 mL/min) or hepatic disease.
11. Abnormal creatine kinase and/or platelet count in the past 6 months (as determined by lab reports obtained from primary care physicians or conducted at baseline).
12. Use of varenicline within the previous 30 days.
13. Ataxia derived from any other cause than genetically-confirmed SCA (including but not limited to alcoholism, head injury, Multiple Sclerosis, olivo-ponto-cerebellar atrophy or multiple system atrophy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Changes in the patient's SARA Rating Scale total score | 25 weeks
Frequency and severity of dose-limiting adverse events | 25 weeks

SECONDARY OUTCOMES:
The effect of varenicline on quality of life in patients with spinocerebellar ataxia | 25 weeks
The effect of varenicline on depression and anxiety ratings | 25 weeks
The effect of varenicline on the activity of daily living (ADL) in patients with spinocerebellar ataxia | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - University of California - Los Angeles, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida